CLINICAL TRIAL: NCT06246773
Title: Feasibility of a Positive Parenting Program for Women Experiencing Homelessness Who Have a History of Interpersonal Violence: A Randomized Controlled Trial
Brief Title: Feasibility of a Positive Parenting Program for Women Experiencing Homelessness Who Have a History of Interpersonal Violence
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Rita and Alex Hillman Foundation - Hillman Emergent Innovation (Unknown)
Responsible Party: Principal Investigator, Doncy Eapen, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-SN-23-1086
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Interpersonal Violence; Homelessness
Keywords: Women experiencing homelessness (WEH); Positive Parenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Parenting Program (Experimental)
  Interventions: Behavioral: Positive Parenting Program
- Usual Care (Active Comparator)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Positive Parenting Program — During the first week, women will receive one session of Recovering from Intimate partner violence through Strengths and Empowerment (RISE) and from week 2 they will receive RISE and PALS simultaneously. Participants will receive four to six components of RISE - education on health effects of violence, improving coping and self-care, enhancing social support, and addressing sexual violence, increase safety planning, and assist in making difficult decisions. During each of the PALS sessions, parents will receive instruction on four responsive parenting constructs: contingent responsiveness, warm sensitivity (responses include high levels of affection and understanding of child states), maintaining vs. redirecting attention to objects and topics of conversation, and verbal scaffolding .In addition to direct instruction, parents will video-record themselves interacting with their child and engage in self-reflection of their own parenting behavior.
  Arms: Positive Parenting Program
Behavioral: Usual Care — Participants will receive services available to them at the shelter or housing facility
  Arms: Usual Care

SUMMARY:
The purpose of this study is to strengthen the skills and self-efficacy of women by addressing the social and emotional trauma that they have experienced from interpersonal violence (IPRV) and homelessness and to promote positive parenting strategies through Play and Learning Strategies (PALS), an evidence based intervention.

ELIGIBILITY:
Inclusion Criteria:

* report of at least one physically violent act from a partner within the past 24 months
* have at least one child 5 years or younger.

Exclusion Criteria:

* do not speak English
* their intimate partner is physically present at the time of enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in Women's parenting stress as assessed by the Parental Stress scale (PSS) | Baseline, immediately after intervention(about 6 weeks after baseline), One month after end of intervention and 3 months after end of intervention intervention
  This is an 18 item questionnaire and each is scored on a 5 point scale from 1(strongly disagree) to (5strongly agree) for a score range of 18-90, higher score indicating more stress
Change in social support as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v 2.0 Emotional Support | Baseline, immediately after intervention(about 6 weeks after baseline), One month after end of intervention and 3 months after end of intervention intervention
  The PROMIS emotional support tool has 16 items and the participants respond each item using a 5-point rating scale from 1(never)-5(always) a higher score indicating more emotional support
Change in social support as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v 2.0 Informational Support | Baseline, immediately after intervention(about 6 weeks after baseline), One month after end of intervention and 3 months after end of intervention intervention
  The PROMIS informational support is a 10 items and participants respond each item using a 5-point rating scale (Health Measures) anchored by 1(never)-5(always) with a higher score indicating a better outcome
Change in women's empowerment as assessed by the Personal Progress Scale-Revised (PPS-R) | Baseline, immediately after intervention(about 6 weeks after baseline), One month after end of intervention and 3 months after end of intervention intervention
  PPS-R is a 28-item self-report measure on which participants rate the extent to which they agreed or disagreed with each item on a 7-point scale.
Change in self efficacy as assessed by the General Self- Efficacy Scale (GSE) | Baseline, immediately after intervention(about 6 weeks after baseline), One month after end of intervention and 3 months after end of intervention intervention
  GSE is a 10 item scale. Participants respond to statements such as "I can solve most problems if I invest the necessary effort" on a 4-point Likert scale anchored by 1(not at all true)-4( exactly true),the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Change in parent satisfaction as assessed by the Parenting Sense of Competence Scale (PSOC) | Baseline, immediately after intervention(about 6 weeks after baseline), One month after end of intervention and 3 months after end of intervention intervention
  The PSOC is a 17-item scale and each item is rated on a 6-point Likert scale anchored by 1(strongly disagree to 6( strongly agree).A higher score indicates a higher parenting sense of competency
Change in children's behavior as assessed by the Devereux Early Childhood Assessments (DECA)-Infant | Baseline, immediately after intervention(about 6 weeks after baseline), One month after end of intervention and 3 months after end of intervention intervention
  DECA (Infant) is a 33 item questionnaire for parents about their infants (1month-18 months) It is a 5 point behavior rating scale scored from never to very frequently which provides an assessment of within-child protective factors central to social and emotional health and resilience.
Change in children's behavior as assessed by the Devereux Early Childhood Assessments (DECA)-Toddler | Baseline, immediately after intervention(about 6 weeks after baseline), One month after end of intervention and 3 months after end of intervention intervention
  DECA (Toddler) is a 36 item questionnaire. It is a 5 point behavior rating scale scored from never to very frequently which provides an assessment of within-child protective factors central to social and emotional health and resilience.
Change in children's behavior as assessed by the Devereux Early Childhood Assessments (DECA)-Preschoolers | Baseline, immediately after intervention(about 6 weeks after baseline), One month after end of intervention and 3 months after end of intervention intervention
  DECA (preschoolers) is a 38 item questionnaire. It is a 5 point behavior rating scale scored from never to very frequently which provides an assessment of within-child protective factors central to social and emotional health and resilience
Change in perceived parent child connectedness as assessed by the Mothers Object Relational Scale- Short Form (MORS- SF) and MORS- Child scale. | Baseline, immediately after intervention(about 6 weeks after baseline), One month after end of intervention and 3 months after end of intervention intervention
  This measures mothers' perception on 2 scales: warmth and invasiveness. This is a 14 item scale and each item is scored from 0( never)-5(always).Warmth is scored by adding the scores from items 1,3,4,6,8,11,and 13, for an average score of 29 a higher score indicating more warmth.
  Invasiveness is scored by adding the scores of items 2,5,7,9,10.12.and 14, an average score of 10 and higher score indicates worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Doncy J Eapen, PhD, MSN, APRN, FNP-BC, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No